CLINICAL TRIAL: NCT05225246
Title: Readmissions After Cardiac Surgical Procedures
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-02023; kt22Reuthebuch
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Cardiac Surgery
Keywords: hospital readmission

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Readmission group: Patients who had heart surgery and returned unplanned to the University Hospital Basel within 30 days of leaving the hospital (outpatient or inpatient)
  Interventions: Other: Data collection on reasons for unplanned readmission to the University Hospital Basel within 30 days of leaving the hospital
- control group: Patients who had heart surgery and did not return unplanned to the University Hospital Basel within 30 days of leaving the hospital (outpatient or inpatient)
  Interventions: Other: Data collection on reasons for unplanned readmission to the University Hospital Basel within 30 days of leaving the hospital

INTERVENTIONS:
Other: Data collection on reasons for unplanned readmission to the University Hospital Basel within 30 days of leaving the hospital — Descriptive analysis of the reasons for unplanned readmissions after cardiac surgery and predictive factors for unplanned readmissions and validation of risk scores

SUMMARY:
The aim of this study is to analyze the reasons for unplanned readmissions after cardiac surgery at the University Hospital Basel. Predictive factors for readmissions and the development over the last 10 years will be analyzed.

ELIGIBILITY:
Inclusion Criteria for readmission group:

* Patients who had heart surgery and returned unplanned to the University Hospital Basel within 30 days of leaving the hospital (outpatient or inpatient)

Inclusion Criteria for control group:

* Patients who had heart surgery and did not return unplanned to the University Hospital Basel within 30 days of leaving the hospital (outpatient or inpatient)

Exclusion Criteria:

* Patients with other initial hospitalization reasons for heart surgery without heart surgery (conservative treatments, cerclage removal, pacemaker surgery) are not included in the analysis.
* Planned readmissions to the University Hospital Basel within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Since January 2010, around 7,500 patients have had heart surgery, and around 2,083 of these patients have returned to the University Hospital of Basel within 30 days of discharge after heart surgery.
Sampling Method: Non-Probability Sample
Enrollment: 4882 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of cardiac related readmissions compared to infections, bleedings and neurological causes | one time assessment at baseline
  Number of cardiac related readmissions compared to infections, bleedings and neurological causes
Sex specific reasons for readmissions | one time assessment at baseline
  Differences in sex specific reasons for readmissions

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Reuthebuch, Prof. Dr. med., Principal Investigator — University Hospital Basel, Cardiac Surgery Clinic
Locations (1):
- University Hospital Basel, Cardiac Surgery Clinic, Basel, Switzerland